CLINICAL TRIAL: NCT02208323
Title: Advancement of Modified Bubble CPAP for the Use in Children in Low Resource Settings: A Study of Safety
Brief Title: Advancement of Modified Bubble CPAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1406M51386; 12985 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Hypoxia; Respiratory Distress
Keywords: Hypoxia; Respiratory Distress
MeSH Terms: conditions — Hypoxia; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bubble CPAP (Experimental): Bubble CPAP for 28 days
  Interventions: Device: Bubble CPAP

INTERVENTIONS:
Device: Bubble CPAP — Respiratory assistance

SUMMARY:
This study proposes that modifying the current form of bCPAP by adjusting the nasal prongs to fit older children, will create a safe form of respiratory support that may help to decrease respiratory distress and thus mortality from pneumonia.

DETAILED DESCRIPTION:
This study proposes that modifying the current form of bCPAP by adjusting the nasal prongs to fit older children, will create a safe form of respiratory support that may help to decrease respiratory distress and thus mortality from pneumonia. Children age 1 month (mo) to 5 years (y) admitted to Gulu Regional Referral Hospital in Gulu, Uganda with respiratory distress will be evaluated for use of the modified bCPAP device as treatment for their respiratory distress (in addition to their routine care, i.e. antibiotics, nutrition support)

ELIGIBILITY:
Inclusion Criteria:

* Age 1mo-5y Hypoxia and/or respiratory distress Hypoxia- Oxygen saturation <92% despite 2LPM nasal cannula support Modified TAL's Respiratory Score >3

Exclusion Criteria:

* Pneumothorax
* Congenital lung disease
* Cyanotic heart disease
* Nasal trauma/facial injury/congenital anomaly (cleft) that makes bubble CPAP nasal interface unusable
* Nasal tissue injury
* Active nosebleed
* Recent abdominal surgery or significant abdominal distension
* Agonal respirations
* GCS <3
* Imminent death within the next 1-2hou

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
determine if a modified bCPAP device with an adapted nasal cannula can be used safely in children outside of the neonatal period | 28 days
  A composite of potential adverse events that could be attributable to bCPAP use. Adverse events such as nasal erosion, nosebleed, and aerophagia will be graded on a scale

SECONDARY OUTCOMES:
show decreased mortality in patients treated with a modified bCPAP respiratory support device. | 28 days
  Comparison of historic mortality data for children admitted with respiratory distress to mortality rate seen during the study. Respiratory distress scores using the TAL score (18) will be recorded prior to therapy and throughout the hospital course

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Bjorklund, MD, Study Director — University of Minnesota
Locations (1):
- Gulu Regional Referral Hospital, Gulu, Uganda

IPD SHARING:
Plan to Share IPD: No